CLINICAL TRIAL: NCT05596656
Title: IgE-mediated Allergies Among Type 1 Diabetes Mellitus Children, Single Centre Observational Study
Status: Completed | Type: Observational
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Engy Osman Ahmed, assistant professor, Mansoura University Children Hospital
Other Study IDs: MS/17.07.21
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Children
MeSH Terms: interventions — Patch Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- allergic type 1 DM children: 45 cases were considered allergic based on written questionnaire taken by the resident. Diagnosis of atopy was confirmed by skin prick testing
  Interventions: Diagnostic Test: skin prick test
- Non-allergic type 1 DM children: Forty-five Non-allergic type 1 DM children were selected as age and sex matched control group.
  Interventions: Diagnostic Test: skin prick test

INTERVENTIONS:
Diagnostic Test: skin prick test — Skin prick testing was performed to all diabetic child with history of allergy. The recommended method of prick testing includes the appropriate use of specific allergen extracts, positive and negative controls, interpretation of the tests after 15 - 20 minutes of application, with a positive result defined as a wheal ≥3 mm diameter more than negative control for detection of specific IgE to one or more of common aeroallergens.
  The location of each allergen was marked with a pen on the volar aspect of forearm to properly identify test results, at least 2 cm from the wrist and the antecubital fossae. The distance between two skin prick tests should be appropriate to avoid false-positive reactions due to direct contamination of a nearby test. A drop of each test solution should be placed on the skin in identical order for each subject tested and immediately pricked with a single-head metal lancet.

SUMMARY:
an interviewer-administrated questionnaire was designed to take history of allergy in diabetic child come to outpatient clinic fulfilling inclusion criteria and used to collect data. Skin prick testing was performed to all diabetic children with history of allergy. Laboratory assessment of Serum Total IgE, IL5 and eosinophils%.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least 2 Years duration of diabetes diagnosed by Criteria for the diagnosis of diabetes mellitus (ISPAD 2018) that include:
* Classic symptoms of diabetes or hyperglycemic crisis, with plasma glucose concentration ≥11.1 mmol/L (200 mg/dL).
* Fasting plasma glucose ≥7.0 mmol/L (≥126 mg/dL). Fasting is defined as no caloric intake for at least 8 hours.
* Two-hour post load glucose ≥11.1 mmol/L (≥200 mg/dL) during an oral glucose tolerance test (OGTT).
* HbA1c ≥6.5%.

Exclusion Criteria:

* presence of other chronic disease associated with DM.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with at least 2 years' duration of Type 1 Diabetes Mellitus. Participants: among 200 cases with Type 1 DM children following up at endocrinology unit
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
positive skin prick test | 20 minutes
  a wheal ≥3 mm diameter more than negative control for detection of specific IgE to one or more of common aeroallergens.

CONTACTS AND LOCATIONS:
Overall Officials: Engy Osman, MD, Study Director — assistant Professor, Pediatrics Department, Faculty of Medicine, Mansoura University, Egypt.
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, None Selected, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinzerling L, Mari A, Bergmann KC, Bresciani M, Burbach G, Darsow U, Durham S, Fokkens W, Gjomarkaj M, Haahtela T, Bom AT, Wohrl S, Maibach H, Lockey R. The skin prick test - European standards. Clin Transl Allergy. 2013 Feb 1;3(1):3. doi: 10.1186/2045-7022-3-3. PMID 23369181